CLINICAL TRIAL: NCT05132842
Title: Determining Patterns of Cannabis Use Among Cancer Patients
Brief Title: Cannabis Use Patterns Among Cancer Patients
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21F.175; P30CA056036-21S3 (NIH); JT 16464 (Other: JeffTrial Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Patients complete a survey about knowledge and awareness of medical cannabis, perceived risks and benefits of cannabis, mode and frequency of use (if applicable), impact on cancer-related symptoms, patient provider discussions about cannabis, and demographic characteristics including health and digital literacy.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete a Survey

SUMMARY:
This study determines patterns of cannabis use among cancer patients. Information collected in this study may help doctors to understand patient use of cannabis therapy, their knowledge and experiences with this therapy, benefits and risks associated with its use, and whether or to what extent they are discussing it with their health care providers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the frequency, modes, and duration of cannabis use, assess experiences with obtaining and using cannabis, as well as reasons for use and perceived risks and benefits of its use among cancer patients who are undergoing or have recently completed active treatment.

Ia. To uncover disparities in use of cannabis, perceptions of use, and communication with providers among cancer patients who are identify as racial and ethnic minorities, have low health or digital literacy, are of older age or low socioeconomic status.

II. Among cancer patients with a known medical marijuana certification, assess the impact of cannabis on pain management, anxiety, anorexia, and quality of life, as well as their communication with their oncology team about their procurement and use of cannabis.

OUTLINE:

Patients complete a survey about knowledge and awareness of medical cannabis, perceived risks and benefits of cannabis, mode and frequency of use (if applicable), impact on cancer-related symptoms, patient provider discussions about cannabis, and demographic characteristics including health and digital literacy.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* English speaking
* Willing to comply with all study procedures and be available for the duration of the study
* Any individual >= 18 years old
* At least one medical or radiation oncology appoint within the last 3 years at one of the SKCC cancer center campuses

Exclusion Criteria:

* Non-English speaking
* Not a cancer patient at one of the SKCC campuses
* Deceased

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had at least one medical or radiation oncology appointment within last 3 years at Sidney Kimmel Cancer Center (SKCC) cancer centers
Sampling Method: Non-Probability Sample
Enrollment: 1568 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Survey data analysis | Up to 12 months
  Respondent demographics and clinical characteristics and survey responses

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States